CLINICAL TRIAL: NCT06244563
Title: Evaluation of the Efficacy of Different Anchorage-supported Appliances and Different Expansion Procedures for Face Mask Treatment in Prepubertal Children
Brief Title: Evaluation of Different Anchorage-supported Appliances and Expansion Procedures for Face Mask Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Gaziantep (Other)
Responsible Party: Principal Investigator, Tugce Ergul, Principal Investigator, University of Gaziantep
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 102
Record Dates: First submitted 2024-01-10; First posted 2024-02-06 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Malocclusion, Angle Class III
Keywords: facemask treatment
MeSH Terms: conditions — Malocclusion, Angle Class III | interventions — Masks

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Face mask with Hybrid-Hyrax and Alt-RAMEC procedure (Experimental): The experimental group was comprised of 15 patients submitted to the alternate rapid maxillary expansion and constriction (alt-RAMEC) procedure for expansion protocol with a hybrid-hyrax expander as anchorage in the maxillary arch. The Face mask was used.
  Interventions: Device: Face mask with Hybrid-Hyrax; Procedure: Alternative Rapid Maxillary Expansion and Contraction Protocol (Alt-RAMEC)
- Face mask with Bonded RME and Alt-RAMEC procedure (Experimental): The experimental group was comprised of 15 patients submitted to the alt-RAMEC procedure for expansion protocol with a bonded RME as anchorage in the maxillary arch. The Face mask was used.
  Interventions: Device: Face mask with Bonded RME; Procedure: Alternative Rapid Maxillary Expansion and Contraction Protocol (Alt-RAMEC)
- Face mask with Hybrid-Hyrax and routine protocol (Experimental): The experimental group was comprised of 15 patients submitted to routine palatal expansion procedure (routine) with a hybrid-hyrax expander as anchorage in the maxillary arch. The Face mask was used.
  Interventions: Device: Face mask with Hybrid-Hyrax; Procedure: Routine Rapid Maxillary Expansion Protocol
- Face mask with Bonded RME and routine protocol (Active Comparator): The active comparator group was comprised of 15 patients who submitted to the routine expansion procedure with a bonded RME as anchorage in the maxillary arch. The Face mask was used.
  Interventions: Device: Face mask with Bonded RME; Procedure: Routine Rapid Maxillary Expansion Protocol

INTERVENTIONS:
Device: Face mask with Hybrid-Hyrax — Participants were treated with face mask using a Hybrid-Hyrax appliance as an anchor in the maxillary arch. The anchorage of hybrid-hyrax appliance was provided by bands adapted to the maxillary first permanent molars and two mini screws in the anterior palate. Force transmission was achieved using intermaxillary elastics that were connected to the face mask arms from the hooks of the hybrid-hyrax appliance in the maxillary canine region.
  Arms: Face mask with Hybrid-Hyrax and Alt-RAMEC procedure; Face mask with Hybrid-Hyrax and routine protocol
Device: Face mask with Bonded RME — Participants were treated with face mask using a bonded RME appliance as an anchor in the maxillary arch. The anchorage of bonded RME appliance was provided by maxillary posterior teeth covered with acrylic cap. Force transmission was achieved using intermaxillary elastics that were connected to the face mask arms from the hooks of the bonded RME in the maxillary canine region.
  Arms: Face mask with Bonded RME and Alt-RAMEC procedure; Face mask with Bonded RME and routine protocol
Procedure: Alternative Rapid Maxillary Expansion and Contraction Protocol (Alt-RAMEC) — In the groups that started with the Alt-Ramec protocol, the parents expanded the appliance screw twice a day in the first week and closed it in the opposite direction in the following week. This process was continued for 7-9 weeks according to the patient's need for expansion.
  Arms: Face mask with Bonded RME and Alt-RAMEC procedure; Face mask with Hybrid-Hyrax and Alt-RAMEC procedure
Procedure: Routine Rapid Maxillary Expansion Protocol — In the groups that started with the routine protocol, parents activated the expansion screw twice a day for 1-2 weeks, depending on the patient's need for expansion.
  Arms: Face mask with Bonded RME and routine protocol; Face mask with Hybrid-Hyrax and routine protocol

SUMMARY:
The purpose of this study is to assess and compare the effect of two appliances (Hybrid-Hyrax expander/ Bonded rapid maxillary expander (RME)) supported by different anchorage units and two different expansion procedures (routine rapid maxillary expansion protocol (routine)/ alternative rapid expansion and constriction protocol (alt-RAMEC)) on maxillary protraction during face mask (FM) treatment.

DETAILED DESCRIPTION:
Face mask therapy is an effective method in the treatment of class III malocclusions due to maxillary insufficiency. In face mask treatment, various intraoral devices are used to transmit protraction forces to the maxilla. According to the anchorage unit, these appliances are divided into tooth-supported and bone-supported. The traditional bonded rapid maxillary expander (RME) is a tooth-supported appliance that allows expansion and is generally used with face masks. However, it causes many side effects due to the transmission of protraction forces through the teeth. Hybrid appliances supported by skeletal and dental anchorage may be preferred over bonded RME in the maxilla for face mask treatment based on their lower dental side effects and high skeletal contribution.

Before transferring the protraction forces to the maxilla using a face mask, expansion is first performed with intraoral devices according to the patient's needs. For this purpose, two different expansion procedures are currently used: routine rapid maxillary expansion (routine) and alternative rapid maxillary expansion and contraction (alt-RAMEC). In the routine rapid maxillary expansion procedure, the expander screw is turned twice a day until the expansion phase is complete. Unlike the routine procedure, in the alt-RAMEC procedure, each week of expansion is followed by a week of contraction. The duration of the expansion-contraction process varies between 7-9 weeks, depending on the patient's need for expansion. These opening and closing phases are increased maxillary protraction by loosening the intermaxillary sutures.

The main purpose of this study is to compare the effects of different combinations of appliances and procedures on maxillary protraction during face mask treatment and determine the most powerful method. Sixty patients who were planned to apply face mask treatment were included in the study and divided into four groups (n=15) (Group 1: Hybrid-Hyrax expander and alt-RAMEC procedure, Group 2: Bonded RME and alt-RAMEC procedure, group 3: Hybrid Hyrax expander and routine protocol, group 4: Bonded RME and routine protocol). To investigate skeletal changes, lateral cephalometric films were taken before (T0) and after (T1) treatment. Dolphin Imaging software and AutoCad 2023 software were used for cephalometric measurements.

ELIGIBILITY:
Inclusion Criteria:

* Skeletal class III
* Prepubertal growth stage
* Reverse overjet

Exclusion Criteria:

* Previous orthodontic treatment history
* Patients with craniofacial abnormalities and syndromes.
* Systemic diseases

Ages: 8 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Actual)
Dates: Start 2022-06-08 (Actual); Primary Completion 2023-04-10 (Actual); Study Completion 2023-06-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of Skeletal and Dental Changes in Millimetric Measurements | 9 month
  Skeletal and dental changes in the maxilla and mandible were evaluated in millimetres using lateral radiographs taken before and after treatment.
  To determine skeletal changes A-VRP (mm), Co-A (mm), A-HRP (mm), Pog-VRP (mm), Co-Gn (mm) and WITS (mm) values were measured.
  To determine dental changes U1-VRP(mm), U1-HRP(mm), U6-VRP(mm), U6-HRP(mm), and L1-VRP(mm) values were measured.

SECONDARY OUTCOMES:
Evaluation of Skeletal and Dental Changes in Angular Measurements | 9 month
  Skeletal and dental changes in the maxilla and mandible were evaluated in angularly using lateral radiographs taken before and after treatment.
  To determine skeletal changes, the following angles were measured: SNA (°), SNB (°), ANB (°), SN-PP (°), SN-MP (°), PP-MP (°) and Ar-Go-Me (°).
  To determine dental changes, the following angles were measured: U1-SN (°) and IMPA (°).

CONTACTS AND LOCATIONS:
Overall Officials: Aysegul Gulec, PhD, Study Chair — University of Gaziantep
Locations (1):
- Gaziantep University, Gaziantep, Sehitkamil, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No